CLINICAL TRIAL: NCT04991532
Title: Research on the Mechanism of Dasatinib Down-regulates the Expression of PD-1 in CMV-activated NKG2C+NK Cells and Enhances Killing pH + Leukemia Stem Cells.
Brief Title: Dasatinib Down-regulates the Expression of PD-1 and Enhances Killing pH + Leukemia Stem Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Dan Xu, professor, Nanfang Hospital, Southern Medical University
Other Study IDs: NFEC-2021-130
Record Dates: First submitted 2021-08-03; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dasatinib group: the CML patient treated with dasatinib
- Imatinib group: the CML patient treated with imatinib

INTERVENTIONS:
Other:

SUMMARY:
Research on the mechanism of dasatinib down-regulates the expression of PD-1 in CMV-activated NKG2C+NK cells and enhances killing pH + leukemia stem cells.

DETAILED DESCRIPTION:
Some patients with CML can withdraw from TKIs after treatment, and the mechanism might be related to the effect of memory NK cells on anti-Ph+ leukemic stem cells (LSCs). Dasatinib affects immune through several pathways including the expression of PD1 in immune cells. Our previous work showed increased NKG2C+ NK cells were found in cases with CMV-DNA+ who suffered Ph+ leukemia and received Dasatinib, and these memory NK cells have anti-LSCs activity. We hypothesize that: CMV infection activates NKG2C+ memory NK cells proliferation; Dasatinib down-regulates the expression of PD1 in PD1+NKG2C+ NK cell subsets and then enhances anti-LSCs activity of these cells. In this study, the effect of Dasatinib on CMV-activated NKG2C+ cell subsets and its mechanism will be studies. Besides, the different NKG2C+ cell subsets on LSCs will be compared. This study might be helpful to clarify the mechanism of TKI withdrawal and to offer foundation for CMV and Ph+ ALL treatment strategies

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old, gender is not limited
2. CML-CP patients treated with TKIs
3. No pregnancy was planned during the treatment

Exclusion Criteria:

1.The researcher judged that it was not suitable to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CML-CP patients treated with TKIs
Sampling Method: Non-Probability Sample
Enrollment: 324 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
NK cells and T cell activation subsets in CML-CP patients treated with TKI for 2 years | 2 years
  NK cells and T cell activation subsets in CML-CP patients treated with TKI for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dan Xu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No